CLINICAL TRIAL: NCT01656161
Title: A Multicentre, Open, Non-comparative, Phase III Study on the Efficacy, Pharmacokinetics, and Safety of Two Subcutaneous Injections of Triptorelin Embonate 22.5 mg 6-month Formulation in Patients With Advanced Prostate Cancer
Brief Title: Study on Efficacy, Pharmacokinetics, and Safety of Two Subcutaneous Injections of Triptorelin Embonate 6 Month Formulation in Patients With Advanced Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Debio 8206-SC-301; KRA75538 (Other: Quintiles)
Record Dates: First submitted 2012-07-31; First posted 2012-08-02 (Estimated); Results first posted 2015-09-15 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triptorelin embonate 22.5 mg (Experimental): Participants received subcutaneous injections of triptorelin embonate 22.5 mg 6-month formulation administered on Day 1 and on Day 169.
  Interventions: Drug: Triptorelin embonate 22.5 mg

INTERVENTIONS:
Drug: Triptorelin embonate 22.5 mg
  Other Names: Pamorelin

SUMMARY:
The primary purpose of this study is to evaluate the efficacy of triptorelin embonate 22.5 mg 6-month formulation administered by the subcutaneous (under the skin) route in:

* achieving castrate levels of testosterone (< 1.735 nmol/L) on Day 29 [i.e., 28 days after investigational medicinal product (IMP) injection], and
* in maintaining serum testosterone castrate levels from Month 2 (Day 57) to end of Month 12 (Day 337) in participants with advanced prostate cancer.

ELIGIBILITY:
Summary Inclusion Criteria:

* Meets protocol-specified criteria for qualification and contraception
* Is willing and able to remain confined in the study unit for the entire duration of each treatment period and comply with restrictions related food, drink and medications
* Voluntarily consents to participate and provides written informed consent prior to any protocol-specific procedures

Summary Exclusion Criteria:

* Has history or current use of over-the-counter medications, dietary supplements, or drugs (including nicotine and alcohol) outside protocol-specified parameters
* Has signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise: 1) the safety or well-being of the participant or study staff; 2) the safety or well-being of the participant's offspring (such as through pregnancy or breast-feeding); 3) the analysis of results

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eija Lundstrom, MD, Study Director — Debiopharm SA; J. Bahlmann, MD, Principal Investigator — Private Practitioner
Locations (10):
- South Africa (10):
  - Paarl Medical Centre, Paarl, Cape Town, Western Cape
  - Vergelegen Medi-Clinic, Somerset West, Cape Town
  - Department of Urology, Tygerberg Hospital, Tygerberg, Cape Town
  - JCM Bahlmann, George, Eastern Cape
  - East Rand Urology Research Unit, Clinix Private Clinic, Johannesburg, Gautang
  - Clinresco Centres (Pty) Ltd, Kempton Park, Gauteng
  - Clinical Trial Unit, Room 2-54, Prinshof Medical Campus, Pretoria, Gauteng
  - Pretoria Urology Hospital, Pretoria, Gauteng
  - Wilmed Park Hospital, Klerksdorp, North West
  - New Groote Schuur Hospital, Division of Urology, Cape Town

REFERENCES:
- [Background] Klippel KF, Winkler CJ, Jocham D, Rubben H, Moser B, Gulati A. [Effectiveness and tolerance of 1 dosage forms (subcutaneous and intramuscular) of decapeptyl depot in patients with advanced prostate carcinoma]. Urologe A. 1999 May;38(3):270-5. doi: 10.1007/s001200050280. German. PMID 10407987
- [Background] Tornoe CW, Agerso H, Senderovitz T, Nielsen HA, Madsen H, Karlsson MO, Jonsson EN. Population pharmacokinetic/pharmacodynamic (PK/PD) modelling of the hypothalamic-pituitary-gonadal axis following treatment with GnRH analogues. Br J Clin Pharmacol. 2007 Jun;63(6):648-64. doi: 10.1111/j.1365-2125.2006.02820.x. Epub 2006 Nov 10. PMID 17096678
- See also: Company website — http://www.debiopharm.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 10 hospital settings in South Africa, from 03 July 2012 to 30 August 2013.
Period: Overall Study
Arm/Group | Triptorelin Embonate 22.5 mg
Started | 120 (Intention to treat analysis set)
Received Triptorelin at Day 1 | 120 (Safety analysis set)
Received Triptorelin at Day 169 | 115
Completed | 113 (Per protocol analysis set)
Not Completed | 7
Not completed — Death | 3
Not completed — Adverse Event | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, defined as all enrolled subjects who received at least one dose of study treatment.
Arm/Group | Triptorelin Embonate 22.5 mg
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.23 (7.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 120
Region of Enrollment [Number; unit: participants]
  South Africa | 120

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving and Maintaining Castrate Levels of Serum Testosterone (<1.735 Nmol/L)
Time Frame: within 337 days
Population: Intention to treat population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Triptorelin Embonate 22.5 mg: Subcutaneous injections of triptorelin embonate 22.5 mg 6-month formulation were administered on Day 1 and on Day 169.
Arm/Group | Triptorelin Embonate 22.5 mg
Number analyzed (Participants) | 120
Percentage of Participants
  Achieving (by Day 29) | 98.33 [94.11 to 99.80]
  Maintaining (Day 57 to Day 337) | 82.61 [74.43 to 89.04]

2. Secondary Outcome: Percentage of Participants Showing ≤ 1.0 IU/L Increase in Serum Luteinising Hormone (LH) From 0 Hour to 2 Hours Post-injection on Day 1 and Day 169
Time Frame: on Days 1 and 169
Population: Intention to treat (ITT) population with a measured value at the time analysed
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Triptorelin Embonate 22.5 mg
Number analyzed (Participants) | 120
percentage of participants
  on Day 1 (n=118) | 0.85 [0.02 to 4.63]
  on Day 169 (n=115) | 87.83 [80.42 to 93.18]

3. Secondary Outcome: Percentage Change From Baseline in Prostate Specific Antigen (PSA) Through Day 337
Time Frame: Baseline through Day 337
Population: ITT population with a measured value at each specified time point
Measure: Mean (Standard Deviation); unit: percentage of change in PSA levels
Arm/Group | Triptorelin Embonate 22.5 mg
Number analyzed (Participants) | 120
percentage of change in PSA levels
  at Day 85 (n=119) | -83.20 (38.10)
  at Day 169 (n=117) | -83.48 (38.29)
  at Day 253 (n=114) | -85.43 (33.94)
  at Day 337 (n=113) | -82.89 (40.74)

4. Secondary Outcome: Number of Participants Who Presented a Real "Acute-on-chronic" (AOC) Phenomenon (Testosterone Levels ≥ 1.735 Nmol/L 48 Hours After the Second Injection While Previously Castrated)
Time Frame: Day 171
Measure: Number; unit: participants
Arm/Group | Triptorelin Embonate 22.5 mg
Number analyzed (Participants) | 120
participants | 1

5. Secondary Outcome: Testosterone Pharmacodynamic (PD) Metrics for First Injection: Area Under the Concentration vs Time Curve (AUC)
Time Frame: Days 1-169
Measure: Geometric Mean (95% Confidence Interval); unit: day*nmol/L
Groups:
- PK/PD Subset: Pharmacokinetic/pharmacodynamic (PK/PD) subset of 15 participants included in the ITT analysis set.
Arm/Group | PK/PD Subset
Number analyzed (Participants) | 15
day*nmol/L | 224.13 [175.82 to 285.72]

6. Secondary Outcome: Testosterone PD Metrics for First Injection: Maximum Concentration (Cmax)
Time Frame: Days 1-169
Measure: Geometric Mean (95% Confidence Interval); unit: nmol/L
Groups:
- PK/PD Subset: PK/PD subset of 15 participants included in the ITT analysis set.
Arm/Group | PK/PD Subset
Number analyzed (Participants) | 15
nmol/L | 16.52 [12.74 to 21.41]

7. Secondary Outcome: Testosterone PD Metrics for First Injection: Time to Peak Serum/Plasma Concentration (Tmax)
Time Frame: Days 1-169
Population: PK/PD subset of 15 participants
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | PK/PD Subset
Number analyzed (Participants) | 15
hours | 48 (40.02) [24 to 48]

8. Secondary Outcome: Testosterone PD Metrics for First Injection: Time to Castration (Tcast)
Time Frame: Days 1-169
Measure: Geometric Mean (95% Confidence Interval); unit: days
Arm/Group | PK/PD Subset
Number analyzed (Participants) | 15
days | 18.01 [16.45 to 19.72]

9. Secondary Outcome: Triptorelin PK Metrics for Both Injections: Area Under the Concentration vs Time Curve (AUC)
Time Frame: Days 1-169 and Days 169-337
Measure: Geometric Mean (95% Confidence Interval); unit: days * ng/mL
Arm/Group | PK/PD Subset
Number analyzed (Participants) | 15
days * ng/mL
  AUC(1-169) | 61.30 [53.50 to 70.25]
  AUC(169-337) | 66.44 [58.99 to 74.82]

10. Secondary Outcome: Triptorelin PK Metrics for Both Injections: Cmax
Time Frame: Days 1-169 and Days 169-337
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Groups:
- PK/PD Subset of 15 Participants: Pharmacokinetic/pharmacodynamic subset of 15 participants who received subcutaneous injections of triptorelin embonate 22.5 mg 6-month formulation administered on Day 1 and on Day 169.
Arm/Group | PK/PD Subset of 15 Participants
Number analyzed (Participants) | 15
ng/mL
  Days 1-169 | 16.77 [13.33 to 21.09]
  Days 169-337 | 18.09 [14.11 to 23.20]

11. Secondary Outcome: Triptorelin PK Metrics for Both Injections: Concentration 0 Hour
Time Frame: Days 1-169 and Days 169-337
Population: Participants in the PK/PD subset with a measured value.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | PK/PD Subset
Number analyzed (Participants) | 12
ng/mL
  Days 1-169 | 0.04 [0.02 to 0.09]
  Days 169-337 | 0.07 [0.04 to 0.11]

ADVERSE EVENTS:
Arm/Group | Triptorelin Embonate 22.5 mg
Serious Adverse Events (participants affected / at risk) | 17/120
Other Adverse Events (participants affected / at risk) | 117/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Triptorelin Embonate 22.5 mg (N=120)
Acute myocardial infarction (Cardiac disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 3
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cystitis (Infections and infestations) | 1
Death (General disorders) | 1
Deep vein thrombosis (Blood and lymphatic system disorders) | 1
Diabetic hyperglycaemic coma (Endocrine disorders) | 1
Femoral neck fracture (Musculoskeletal and connective tissue disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Hip fracture (Musculoskeletal and connective tissue disorders) | 1
Hyperglycaemia (Endocrine disorders) | 2
Hypersensitivity (Immune system disorders) | 1
Meningitis streptococcal (Infections and infestations) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 2
Paraparesis (Nervous system disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Radius fracture (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Triptorelin Embonate 22.5 mg (N=120)
Constipation (Gastrointestinal disorders) | 11
Lethargy (General disorders) | 11
Upper respiratory tract infection (Infections and infestations) | 8
Urinary tract infection (Infections and infestations) | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Back pain (Musculoskeletal and connective tissue disorders) | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 6
Erectile dysfunction (Reproductive system and breast disorders) | 10
Hot flush (Vascular disorders) | 86
Hypertension (Vascular disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreement restricts the PI from discussing or publishing trial results after the trial is completed.